CLINICAL TRIAL: NCT01045460
Title: Randomized Trial of Activated Marrow Infiltrating Lymphocytes Alone or in Conjunction With an Allogeneic GM-CSF-based Myeloma Cellular Vaccine in the Autologous Transplant Setting in Multiple Myeloma
Brief Title: Trial of Activated Marrow Infiltrating Lymphocytes Alone or in Conjunction With an Allogeneic Granulocyte Macrophage Colony-stimulating Factor (GM-CSF)-Based Myeloma Cellular Vaccine in the Autologous Transplant Setting in Multiple Myeloma
Acronym: aMILs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0997; NA_00029491 (Other: JHMIRB)
Record Dates: First submitted 2009-12-14; First posted 2010-01-11 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — N(1)-methyl-2-lysergic acid diethylamide; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Leukapheresis; Blood Component Removal; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASCT + MILs (Experimental): Cyclophosphamide and filgrastim will be given to mobilize peripheral blood stem cells. Leukapheresis will be performed to collect peripheral blood from which activated marrow infiltrating lymphocytes will be produced. A melphalan conditioning regimen will be used prior to autologous stem cell transplant, and the MILs product will be administered on Days 3 and 4.
  Interventions: Biological: Activated marrow infiltrating lymphocytes; Drug: Cyclophosphamide; Biological: Filgrastim; Procedure: Leukapheresis; Drug: Melphalan; Biological: Autologous stem cell transplant
- ASCT + MILs + vaccine (Experimental): Cyclophosphamide and filgrastim will be given to mobilize peripheral blood stem cells. Leukapheresis will be performed to collect peripheral blood from which activated marrow infiltrating lymphocytes will be produced. A melphalan conditioning regimen will be used prior to autologous stem cell transplant, and the MILs product will be administered on Days 3 and 4. The allogeneic myeloma vaccine will be administered on Days 21, 60, 180, and 300.
  Interventions: Biological: Activated marrow infiltrating lymphocytes; Biological: Allogeneic Myeloma Vaccine; Drug: Cyclophosphamide; Biological: Filgrastim; Procedure: Leukapheresis; Drug: Melphalan; Biological: Autologous stem cell transplant

INTERVENTIONS:
Biological: Activated marrow infiltrating lymphocytes — Administered on Days 3 and 4.
  Other Names: MILs; aMILs
Biological: Allogeneic Myeloma Vaccine — Allogeneic granulocyte macrophage colony-stimulating factor (GM-CSF)-based myeloma cellular vaccine. Administered on Days 21, 60, 180, and 300.
  Arms: ASCT + MILs + vaccine
Drug: Cyclophosphamide — Administered at 2.5 g/m^2.
  Other Names: Cytoxan
Biological: Filgrastim — Administered post cyclophosphamide daily until leukapheresis.
  Other Names: G-CSF
Procedure: Leukapheresis — Performed approximately 12 days post cyclophosphamide. Exact date depends on peripheral blood CD34+ cell counts.
  Other Names: Apheresis
Drug: Melphalan — 100 mg/m^2/day given on Days -2 and -1.
  Other Names: Alkeran
Biological: Autologous stem cell transplant — Infused on Day 0.
  Other Names: ASCT

SUMMARY:
Patient Population: Patients with active myeloma (Stage II/III) that have completed induction therapy and are eligible for an autologous stem cell transplant.

Number of Patients: Will treat a total of 32 evaluable patients in a 1:1 randomization of aMILs vs aMILs plus vaccine. An evaluable patient is defined as one which has received the activated MILs and is at least 6 months post-transplant.

Study Objectives:

Disease response as determined by the Blade' criteria will be the primary endpoint of the trial at one year.

Additional study endpoints include progression free survival, parameters of T cell reconstitution, anti-tumor immune responses as well as the effect on osteoclastogenesis and clonogenic myeloma precursor cells.

ELIGIBILITY:
Inclusion Criteria:

* Durie-Salmon Stage II or III multiple myeloma
* Newly diagnosed either prior to receiving treatment or having completed induction therapy
* Relapsed myeloma not previously transplanted within the past 5 years
* Measurable serum and/or urine M-protein from prior to induction therapy documented and available. A positive serum free lite assay is acceptable
* Age greater than 18 years old
* ECOG performance status of 0 - 2
* Meet all institutional requirements for autologous stem cell transplantation
* The patient must be able to comprehend and have signed the informed consent

Exclusion Criteria:

* Diagnosis of any of the following plasma cell disorders: POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein] and skin changes) Non-secretory myeloma (no measurable protein on Serum Free Lite Assay)
* Plasma cell leukemia
* Amyloidosis
* Use of corticosteroids (glucocorticoids) within 21 days of pre-transplant vaccine or bone marrow collection
* Use of any myeloma-specific therapy other than lenalidomide within 21 days of pre-transplant vaccine
* In a complete remission at the time of bone marrow collection
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within seven days of vaccination or bone marrow collection
* Participation in any clinical trial, within four weeks prior to vaccination or bone marrow collection on this trial, which involved an investigational drug or device
* History of malignancy other than multiple myeloma within five years of vaccination or bone marrow collection, except adequately treated basal or squamous cell skin cancer
* Active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis) requiring systemic treatment. Hypothyroidism without evidence of Grave's Disease or Hashimoto's thyroiditis is permitted
* Evidence of spinal cord compression at time of transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01-15 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borrello, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was a screen failure.
Groups:
- ASCT + MILs + Vaccine: Cyclophosphamide and filgrastim will be given to mobilize peripheral blood stem cells. Leukapheresis will be performed to collect peripheral blood from which activated marrow infiltrating lymphocytes will be produced. A melphalan conditioning regimen will be used prior to autologous stem cell transplant, and the MILs product will be administered on Days 3 and 4. The allogeneic myeloma vaccine will be administered on Days 21, 60, 180, and 300.
  Activated marrow infiltrating lymphocytes: Administered on Days 3 and 4.
  Allogeneic Myeloma Vaccine: Allogeneic granulocyte macrophage colony-stimulating factor (GM-CSF)-based myeloma cellular vaccine. Administered on Days 21, 60, 180, and 300.
  Cyclophosphamide: Administered at 2.5 g/m^2.
  Filgrastim: Administered post cyclophosphamide daily until leukapheresis.
  Leukapheresis: Performed approximately 12 days post cyclophosphamide. Exact date depends on peripheral blood CD34+ cell counts.
  Melphalan: 100 mg/m^2/day given on Days -2
Period: Overall Study
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Started | 17 | 18
Completed | 11 | 15
Not Completed | 6 | 3
Not completed — Physician Decision | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 6 | 7 | 13
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 69] | 63 [39 to 72] | 60 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
International Staging System (ISS) stage [Count of Participants; unit: Participants] — * Stage 1: Beta-2 microglobulin < 3.5 mg/L and serum albumin >= 3.5 g/dL.
  * Stage 2: Neither stage 1 nor stage 3.
  * Stage 3: Beta-2 microglobulin >= 5.5 mg/L.
  Higher beta-2 microglobulin reflects greater tumor mass. Therefore, a higher stage reflects a worse prognosis.
  Participants
    Stage 1 | 7 | 8 | 15
    Stage 2 | 3 | 4 | 7
    Stage 3 | 3 | 5 | 8
    Stage unknown | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rates by Blade Criteria
Description: Number of participants with each disease response category utilizing the Blade criteria:
  * Complete Response (CR): Defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
  * Near Complete Response (nCR): Defined as negative serum and urine paraprotein, positive serum and/or urine immunofixation, and a bone marrow aspirate with < 5% plasma cells.
  * Very Good Partial Response (VGPR): Defined as negative serum and urine paraprotein with positive serum and/or urine immunofixation; or a 90% decrease in serum paraprotein with urine paraprotein < 100 mg/24 hours.
  * Partial Response (PR): Defined as a 50-89% decrease in serum paraprotein.
  * Minimal Response (MR): Defined as a 25-49% decrease in serum paraprotein.
  * Stable Disease (SD): Defined as not falling into any other response category.
  * Overall response rate (ORR): Total of CR, nCR, VGPR, and PR.
Time Frame: Up to 1 year
Population: Only participants who had ASCT were evaluated for response. Three participants on the ASCT + MILs arm and two participants on the ASCT + MILs + vaccine arm were removed from study prior to ASCT and were therefore not evaluable for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 14 | 16
Participants
  CR | 2 | 5
  nCR | 3 | 2
  VGPR | 1 | 1
  PR | 4 | 5
  MR | 0 | 1
  SD | 4 | 2
  ORR | 10 | 13

2. Secondary Outcome: Progression-free Survival
Description: Median number of months that participants were alive without disease relapse or progression (progression-free survival).
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 14 | 16
months | 15.5 [13 to 37] | 18.6 [13 to 27]

3. Secondary Outcome: Overall Survival
Description: Number of participants alive at 5 years (overall survival).
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 14 | 16
Participants | 7 | 9

4. Secondary Outcome: Feasibility as Measured by Participant Withdrawal or Removal
Description: Number of participants who withdrew or were removed from the study for reasons other than lack of efficacy prior to completion.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 17 | 18
Participants | 3 | 3

5. Secondary Outcome: Safety as Measured by Grade 3-5 Adverse Events
Description: Number of participants who experienced at least one grade 3-5 adverse event by CTCAE 3.0 that was attributed to MILs or the myeloma vaccine.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 17 | 18
Participants | 0 | 1

6. Secondary Outcome: Anti-tumor Immune Response
Description: * Evaluate tumor specific responses in blood and bone marrow
  * Examine T cell responses to DC-pulsed myeloma cell lines
  * Examine induction of novel antibody responses
Time Frame: Days 60, 180, and 360
Population: This measure was not assessed. Data was not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: The Effect of aMILs on Osteoclastogenesis as Measured by Bone Turnover (RANKL/OPG Ratio)
Time Frame: Days 60, 180, and 360
Population: This measure was not assessed. Data was not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: The Effect of aMILs on Osteoclastogenesis as Measured by Bone Turnover (Serum C Telopeptide Levels)
Description: Serum C Telopeptide
Time Frame: Days 60, 180, 360
Population: This measure was not assessed. Data was not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: The Effect of aMILs on Osteoclastogenesis as Measured by Bone Turnover (bAlkaline Phosphatase Levels)
Description: bAlkaline phosphatase
Time Frame: Days 60, 180, 360
Population: This measure was not assessed. Data was not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: The Effect of aMILs on Osteoclastogenesis as Measured by Bone Turnover (Osteocalcin Levels)
Description: Osteocalcin
Time Frame: Days 60, 180, 360
Population: This measure was not assessed. Data was not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Effect of aMILs on Clonogenic Myeloma Precursors
Description: • Examine side population of CD19 enriched PBLs throughout study.
Time Frame: Days 60, 180, and 360
Population: This measure was not assessed. Data was not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: All adverse events related to MILs or vaccine administration were collected. Adverse events related to ASCT were not collected.
Arm/Group | ASCT + MILs | ASCT + MILs + Vaccine
All-Cause Mortality (participants affected / at risk) | 7/17 | 6/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 6/17 | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASCT + MILs (N=17) | ASCT + MILs + Vaccine (N=18)
Anemia (Investigations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Fever (Immune system disorders) | 0 (0) | 1 (1)
Flu-like symptoms (Immune system disorders) | 0 (0) | 1 (1)
Injection site reaction (Immune system disorders) | 0 (0) | 14 (40)
Pancytopenia (Investigations) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-08-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT01045460/Prot_SAP_000.pdf